CLINICAL TRIAL: NCT07070128
Title: Screening Tool Artificial Intelligence-based for Predicting the Genetic Risk of BREAST Cancer (STAR-BREAST)
Brief Title: Screening Tool Artificial Intelligence-based for Predicting the Genetic Risk of BREAST Cancer
Acronym: STAR-BREAST
Status: Recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D0817R00113
Record Dates: First submitted 2025-04-16; First posted 2025-07-17 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Breast Neoplasms
Keywords: Breast Cancer; Artificial Intelligence; Genetic Risk
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

SUMMARY:
It is a retrospective observational study that will include female patients aged 18 years or older, who were treated between 2017 and 2024, in both public and private institutions, and identified as at high genetic risk by breast specialists and referred to a geneticist. The artificial intelligence-based tool to be used in this study is developed by the startup WeConecta, which will collect data via WhatsApp about the patients' family cancer history with the aim of predicting the genetic risk of developing breast cancer.

DETAILED DESCRIPTION:
This is an observational retrospective study. Patients considered by mastologists to be at genetic risk and who have undergone genetic testing with a geneticist will have their electronic medical records reviewed and, if eligible for the study, will answer questions conducted by the virtual assistant using AI about their family history of cancer.

This study will be conducted in two centers. The first is the Breast Center at Hospital Moinhos de Vento, designated as the coordinating center, located in Porto Alegre, Rio Grande do Sul, Brazil. It is a private center composed of a multidisciplinary team dedicated to breast health care, from routine exams for early detection of malignant tumors, diagnosis, comprehensive treatment at different stages of the disease, to post-treatment follow-up. The second center, designated as a participant, is the Human Genetics Center (CEGH/ICB), located in Goiânia, Brazil. This entity works interdisciplinarily and is linked to the Institute of Biological Sciences at the Federal University of Goiás (UFG), with the aim of developing activities in diagnosis, education, research, and outreach in the field of human genetics.

CEGH/ICB is a public institution that serves women with breast cancer from the Unified Health System (SUS), and its role in the research is to share collected data from the population of interest with the coordinating center.

ELIGIBILITY:
Inclusion Criteria:

* female patients,
* aged 18 years or older,
* identified as high genetic risk by breast surgeons,
* referred to a geneticist, and
* who agree to participate in the study.

Exclusion Criteria:

* male patients,
* absence of complete information in the medical records,
* patients unaware of their biological family history, and
* patients who do not agree to participate in the study.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Convenience sampling will be performed, inviting all women treated at both institutions from January 2017 to June 2024 who have been considered by breast surgeons as genetic risk patients and have undergone genetic testing with a geneticist, regardless of whether they have invasive breast carcinoma.
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2025-08-20 (Actual); Primary Completion 2026-08-11 (Estimated); Study Completion 2026-08-11 (Estimated)

PRIMARY OUTCOMES:
Agreement between AI tool results and genetic test results | Through study completion, an average at one year.
  Implement the use of an artificial intelligence (AI)-based tool, WeConecta, to predict the genetic risk of hereditary breast cancer in women treated at a private and public institution, including analyses of the sensitivity, specificity, and positive and negative predictive values of the tool in comparison with the results of the genetic test. Hypothesis: The artificial intelligence (AI)-based tool may present a strong level of agreement regarding the indication for genetic counseling in relation to the indication of mastologists, impacting genetic testing.

SECONDARY OUTCOMES:
Evaluate the rate of agreement between the AI tool and the breast surgeon | Through study completion, an average at one year.
  Comparison between the number of participants who were indicated to genetic counseling through the AI tool and according to the opinion of the mastologist
Agreement between hereditary breast cancer risk identified by the AI tool and the results of genetic testing. | Through study completion, an average at one year.
  To assess how many patients were identified by the AI tool as having "hereditary breast cancer risk" and how closely they agreed with the actual number obtained from genetic testing results.
Describe the rate of family history profile of women at high risk for breast cancer | Through study completion, an average at one year.
  Describe the rate of family history profile of women at high risk for breast cancer
Examine the rate of high penetrance variants | Through study completion, an average at one year.
  Examine the rate of high penetrance variants.
Describe the rate of profile of patients with confirmed BRCA1 and BRCA2 variants | Through study completion, an average at one year.
  Describe the rate of profile of patients with confirmed BRCA1 and BRCA2 variants
Compare the rate of patient profiles between the two institutions | Through study completion, an average at one year.
  Compare the rate of patients with pathogenic variants and genetic risk of breast cancer between the two institutions involved in the study.

CONTACTS AND LOCATIONS:
Locations (2):
- Brazil (2):
  - Research Site, Golania, Goiás
  - Research Site, Porto Alegre, Rio Grande do Sul

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/